CLINICAL TRIAL: NCT02824419
Title: Imaging of Active Granulomas With [18F]FDG and Selected Inflammatory PET Tracers in Pulmonary Sarcoidosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: T16/2015
Record Dates: First submitted 2016-05-27; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — Methionine; 68Ga-DOTANOC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- C11-methionine (Experimental): To compare FDG and C11-methionine in the detection of sarcoidotic lesions.
  Interventions: Drug: Methionine
- 68Ga-Dotanoc (Experimental): To compare FDG and 68Ga-DOTANOC in the detection of sarcoidotic lesions.
  Interventions: Drug: DOTANOC

INTERVENTIONS:
Drug: Methionine — Subject undergoes imaging studies with FDG and with methionine.
  Other Names: PET tracers
  Arms: C11-methionine
Drug: DOTANOC — Subject undergoes imaging studies with FDG and with DOTANOC.
  Other Names: PET tracers
  Arms: 68Ga-Dotanoc

SUMMARY:
The goal of the current study is to evaluate the potential of the selected PET tracers to detect sarcoidotic lesions in lungs. The tracers are already in clinical use for the detection of certain inflammatory processes or malignant tumors, and their targets present similarities with molecular mechanisms of sarcoidosis.

DETAILED DESCRIPTION:
The diagnosis of sarcoidosis is difficult since there is no specific noninvasive method available to diagnose sarcoidosis. FDG-PET imaging is in use, however, FDG is not a specific tracer for sarcoidosis and other inflammatory diseases may interfere with the imaging findings. The aim of the current protocol is to evaluate the potential of other inflammatory PET-tracers in the detection of sarcoidotic lesions.

The patients with active sarcoidotic lesions in lungs will be recruited. First, the patient undergoes PET-FDG scan and then the patient undergoes the PET scan either with C11-methionine or 68Ga-DOTANOC. The results with the latter tracers will be compared to the imaging results with FDG.

ELIGIBILITY:
Inclusion Criteria:

* Patient with sarcoidosis

Exclusion Criteria:

* any malignant disease
* any significant other inflammatory or infectious disease affecting lungs
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The detection of sarcoidotic lesion with C11-methionine or 68Ga-DOTANOC. | baseline
  Qualitative assessment of tracer uptake in sarcoidotic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Knuuti, MD, PhD, Principal Investigator — Turku PET Centre, Turku University Hospital, Turku, Finland
Locations (1):
- Turku University Hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No